CLINICAL TRIAL: NCT04336215
Title: Cohort Study of SARS-CoV-2 Incidence, Transmission, and Disease Severity in Healthcare Workers
Brief Title: Rutgers COVID-19 Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Reynold Panettieri, MD, Director, Rutgers Institute for Translational Medicine & Science, Rutgers, The State University of New Jersey
Other Study IDs: 2020000679
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Coronavirus; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasopharyngeal or throat swabs, saliva, and blood (for detecting SARS-CoV-2 positivity and immunity)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthcare Workers: 546 HCW with high intensity direct patient care from two RBHS-affiliated academic hospitals: Robert Wood Johnson University Hospital (New Brunswick, NJ) and University Hospital (Newark, NJ) and Rutgers School of Dental Medicine (Newark, NJ).
  Interventions: Other: Non-Interventional
- Non-Healthcare Workers: 283 non-healthcare workers (NHCW) from Rutgers faculty, postdoctoral students, students, other trainees, administrators, and staff who do not have patient contact.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — This non-interventional study poses no additional risks to people with pre-existing conditions.

SUMMARY:
Our long-term goal is to protect the health care workforce (HCW) caring for SARS-CoV-2-infected patients, their families, communities, and the general population. Our specific objective is to rapidly establish a prospective cohort to characterize the factors related to viral transmission and disease severity in a large healthcare system. We addressed this hypothesis by recruiting and longitudinally following 546 HCW and a comparison group of 283 non-HCW within a large academic health system, Rutgers Biomedical and Health Sciences (RBHS). By intensively following participants over a several year period (2020-2024) and collecting serial biospecimens (nasopharyngeal/throat swabs, blood, and saliva) and questionnaire data at multiple time points, we will uniquely characterize SARS-CoV-2 transmission and risk factors for COVID-19 among HCW and our larger academic community.

DETAILED DESCRIPTION:
This prospective longitudinal cohort study is comprised of: (1) 546 HCW from two RBHS hospitals: Robert Wood Johnson University Hospital (RWJUH) in New Brunswick and University Hospital (UH) in Newark ; (both hospital presidents have approved the study) (2) 283 NHCW from Rutgers faculty, staff, and hospital employees without patient contact. At baseline, investigators will obtain nasopharyngeal or throat swabs, saliva, and blood (for detecting SARS-CoV-2 positivity and immunity, respectively) and collect questionnaire data on sociodemographic factors, lifestyle, and medical history. In the first phase of the study, nasopharyngeal/throat swabs, saliva, and blood collection were collected every two weeks for two months, after which monthly samples were collected for four additional months (9 visits total, including baseline). Weekly questionnaire data and daily temperature data was collected from each participant for the first two months of the study. Investigators will calculate and compare incidence rates and risk factors of SARS-CoV-2 positivity and COVID-19 in healthcare workers and non-healthcare workers and assess symptoms and severity of disease. Through additional funding, we will continue to administer follow-up questionnaires and collect additional specimens (primarily for serology) through 2024.

Our specific aims are:

1. To assess the baseline prevalence of SARS-CoV-2 and COVID-19 in the study population.
2. To characterize the natural history of SARS-CoV-2 infection in a diverse US workforce, including the incidence of asymptomatic infections and critical illness.
3. To determine the incidence of SARS-CoV-2 and COVID-19 in healthcare workers compared with non-healthcare workers.
4. To identify the risk factors for acquiring SARS-CoV-2 and developing COVID-19.
5. To determine the duration and extent of SARS-CoV-2 shedding.
6. To determine immune responses to SARS-CoV-2 infection and or vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* 20 years and older
* Hospital and RBHS healthcare workers who have regular direct patient contact (≥3 patients/shift) in emergency rooms or inpatient settings that is expected to continue regularly over the next ≥3 months and who work ≥20 hours in the hospital weekly (residents, clinical fellows, attending physicians, nurse practitioners, physician assistants, registered nurses, license practice nurses, medical technicians, respiratory therapists, physical therapists, clinical pharmacists, dentists, dental hygienists, or dental assistants)
* Hospital workers who do not have patient contact and non-healthcare from the Rutgers faculty, postdoctoral students, administrators, and staff.

Exclusion Criteria:

* Previous diagnosis with COVID-19
* Pregnant or have been diagnosed with a new medical condition in the past 30 days or have had a change in medications in the past 30 days
* Participants who have been hospitalized in the past 30 days, had and had an emergency room, urgent care visit, or have had surgery.
* Participants who have a fever on the day of their first visit to the study site (for consent, biospecimen collection, etc.).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * HCW from two RBHS hospitals: Robert Wood Johnson University Hospital (RWJUH) in New Brunswick and University Hospital (UH) in Newark ; (both hospital presidents have approved the study)
  * NHCW from Rutgers faculty, staff, and hospital employees without patient contact;
Sampling Method: Non-Probability Sample
Enrollment: 829 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence | up to 24 weeks
  Prevalence and 95% confidence intervals, using standard epidemiological methods (Aims 1, 2, and 3).
Incidence | up to 24 weeks
  Incidence and 95% confidence intervals, using standard epidemiological methods (Aims 1, 2, and 3).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Carson, MD, Principal Investigator — Rutgers Biomedical Health Sciences; Reynold A Panettieri, MD, Principal Investigator — Rutgers Institute for Translational Medicine and Science
Locations (7):
- United States (7):
  - Clinical Research Center Rutgers-Robert Wood Johnson Medical School RWJUH East Tower -, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Clinical Research Unit Rutgers New Jersey Medical School, Newark, New Jersey
  - Rutgers School of Dental Medicine, Newark, New Jersey
  - University Hospital, Newark, New Jersey
  - Environmental and Occupational Health Sciences Institute, Piscataway, New Jersey
  - RUCDR Infinite Biologics, Piscataway, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colizza V, Barrat A, Barthelemy M, Valleron AJ, Vespignani A. Modeling the worldwide spread of pandemic influenza: baseline case and containment interventions. PLoS Med. 2007 Jan;4(1):e13. doi: 10.1371/journal.pmed.0040013. PMID 17253899
- [Background] Bai Y, Yao L, Wei T, Tian F, Jin DY, Chen L, Wang M. Presumed Asymptomatic Carrier Transmission of COVID-19. JAMA. 2020 Apr 14;323(14):1406-1407. doi: 10.1001/jama.2020.2565. PMID 32083643
- [Background] Schulert GS, Zhang M, Fall N, Husami A, Kissell D, Hanosh A, Zhang K, Davis K, Jentzen JM, Napolitano L, Siddiqui J, Smith LB, Harms PW, Grom AA, Cron RQ. Whole-Exome Sequencing Reveals Mutations in Genes Linked to Hemophagocytic Lymphohistiocytosis and Macrophage Activation Syndrome in Fatal Cases of H1N1 Influenza. J Infect Dis. 2016 Apr 1;213(7):1180-8. doi: 10.1093/infdis/jiv550. Epub 2015 Nov 23. PMID 26597256
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Mahase E. Covid-19: WHO declares pandemic because of "alarming levels" of spread, severity, and inaction. BMJ. 2020 Mar 12;368:m1036. doi: 10.1136/bmj.m1036. No abstract available. PMID 32165426
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Han Y, Yang H. The transmission and diagnosis of 2019 novel coronavirus infection disease (COVID-19): A Chinese perspective. J Med Virol. 2020 Jun;92(6):639-644. doi: 10.1002/jmv.25749. Epub 2020 Mar 12. PMID 32141619
- [Background] Anderson RM, Heesterbeek H, Klinkenberg D, Hollingsworth TD. How will country-based mitigation measures influence the course of the COVID-19 epidemic? Lancet. 2020 Mar 21;395(10228):931-934. doi: 10.1016/S0140-6736(20)30567-5. Epub 2020 Mar 9. No abstract available. PMID 32164834
- [Background] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- [Background] Fauci AS, Lane HC, Redfield RR. Covid-19 - Navigating the Uncharted. N Engl J Med. 2020 Mar 26;382(13):1268-1269. doi: 10.1056/NEJMe2002387. Epub 2020 Feb 28. No abstract available. PMID 32109011
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Pan X, Chen D, Xia Y, Wu X, Li T, Ou X, Zhou L, Liu J. Asymptomatic cases in a family cluster with SARS-CoV-2 infection. Lancet Infect Dis. 2020 Apr;20(4):410-411. doi: 10.1016/S1473-3099(20)30114-6. Epub 2020 Feb 19. No abstract available. PMID 32087116
- [Background] Del Rio C, Malani PN. COVID-19-New Insights on a Rapidly Changing Epidemic. JAMA. 2020 Apr 14;323(14):1339-1340. doi: 10.1001/jama.2020.3072. No abstract available. PMID 32108857
- [Background] Zhang H, Penninger JM, Li Y, Zhong N, Slutsky AS. Angiotensin-converting enzyme 2 (ACE2) as a SARS-CoV-2 receptor: molecular mechanisms and potential therapeutic target. Intensive Care Med. 2020 Apr;46(4):586-590. doi: 10.1007/s00134-020-05985-9. Epub 2020 Mar 3. No abstract available. PMID 32125455
- [Derived] Horton DB, Barrett ES, Roy J, Gennaro ML, Andrews T, Greenberg P, Bruiners N, Datta P, Ukey R, Velusamy SK, Fine D, Honnen WJ, Yin YS, Pinter A, Brooks A, Tischfield J, Hussain S, Jagpal S, Swaminathan S, Parmar V, Reilly N, Gaur S, Panettieri RA, Carson JL, Blaser MJ. Determinants and Dynamics of SARS-CoV-2 Infection in a Diverse Population: 6-Month Evaluation of a Prospective Cohort Study. J Infect Dis. 2021 Oct 28;224(8):1345-1356. doi: 10.1093/infdis/jiab411. PMID 34387310